CLINICAL TRIAL: NCT03890302
Title: A Phase 1, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of Single and Multiple Ascending Doses of FB704A
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics,and Clinical Activity of FB704A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fountain Biopharma Inc. (Industry)
Collaborators: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: FB704ACLIS-01-RA
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A (Experimental): 0.5 mg/kg study drug, or placebo, administered once
  Interventions: Drug: FB704A; Drug: Placebo
- Cohort B (Experimental): 2 mg/kg study drug, or placebo, administered once
  Interventions: Drug: FB704A; Drug: Placebo
- Cohort C (Experimental): 4 mg/kg study drug, or placebo, administered once
  Interventions: Drug: FB704A; Drug: Placebo
- Cohort D (Experimental): 8 mg/kg study drug, or placebo, administered once
  Interventions: Drug: FB704A; Drug: Placebo
- Cohort E (Experimental): Starting dose of 2 mg/kg or approximately half the maximum tolerated dose (MTD) in Part 1 (Cohorts A-D), whichever is lower, up to 4 mg/kg; or placebo. Administered 4 times (approximately once every 2 weeks).
  Interventions: Drug: FB704A; Drug: Placebo

INTERVENTIONS:
Drug: FB704A — Administered by IV infusion
Drug: Placebo — Identical in appearance and same excipients as FB704A, but without active compound. Administered by IV infusion

SUMMARY:
The cause of Rheumatoid Arthritis (RA) is not fully understood. However, one of the substances secreted by certain cells in the body, interleukin-6 (IL-6), is believed to play a major role in chronic inflammation that is typical in RA. This study investigates the drug FB704A, which is believed to lower the inflammation caused by IL-6. This study will be in 2 sequential parts: a single increasing dose part (Part 1) and a multiple-increasing dose part (Part 2). Subjects will receive either active or placebo drug by IV infusion. Subjects in both parts will have a short stay in the clinic at the start of the study, then will return for outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent.
* No significant clinical, cardiac or physical abnormalities (Part 1 of study).
* Diagnosis of Rheumatoid Arthritis as defined by 2010 revised American College of Rheumatology (ACR) more than 3 months prior to start of study (Part 2 of study).
* If using oral corticosteroids (prednisone ≤ 10mg or equivalent) and/or NSAIDS, subjects must be on stable dose(s) for at least 14 days prior to start of Part 2 of study and dose must be expected to remain stable through end of Part 2 of study.
* Subjects must be being treated with 1 or a combination of disease modifying antirheumatic drugs (DMARDs) methotrexate, leflunomide, sulfasalazine, and/or hydroxychloroquine (but not simultaneous use of leflunomide and methotrexate), at any dose for at least 28 days prior to start of Part 2 of study and on a stable dose(s) for at least 14 days prior to start of Part 2 of study.
* Subjects with documented RA that meet all inclusion criteria but are not taking DMARDs may be permitted in Part 2 of the study at the discretion of an investigator.
* Women of childbearing potential must agree to use one of the accepted contraceptive regimens from at least 30 days prior to first administration of the study medication, during the study, and for at least 60 days after last dose of the study medication.
* Women of non-childbearing potential should be surgically sterile or in a menopausal state (at least 1 year without menses).
* All males must agree to use highly effective contraception and to not donate sperm throughout the study and for 90 days following last dose of study medication.
* Subjects must have a body weight ≥ 50 kg at screening and a body mass index (BMI) of 19.0 to 30.0 kg/m2, inclusive (Part 2 of study).
* Subjects must have not smoked or used any nicotine products for at least 3 months before screening (Part 1 of study).

Exclusion Criteria:

* Women who are pregnant or lactating.
* Subject has a past history of, or a history of risk factors for, heart arrhythmias or long QT syndrome.
* Subject has recurrent chronic serious infection, or has had a serious infection within 60 days of start of study.
* Subject has latent or active tuberculosis.
* Subject has received any live attenuated vaccine (e.g. varicella-zoster, oral polio, rabies, flu vaccine) within 3 months of start of study.
* Subject has received any biological drug or blood product within 3 months or 5 half-lives of start of study; or has received any other study drug within 30 days or 5 half-lives of start of study.
* Subject has previously been treated with any biologic, anti-interleukin-6 (anti-IL-6) or interleukin-6 receptor (IL-6) antagonist and/or has previous exposure to the study drug.
* Subjects with a documented history of an autoimmune disease other than rheumatoid arthritis or secondary Sjogren's syndrome.

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) (Part 1) | Up to Day 57
Incidence of Adverse Events (AEs) (Part 2) | Up to Day 99
Number of participants with clinical laboratory abnormalities (Part 1) | Up to Day 57
Number of participants with clinical laboratory abnormalities (Part 1) | Up to Day 99
Number of participants with physical examination abnormalities (Part 1) | Up to Day 57
Number of participants with physical examination abnormalities (Part 2) | Up to Day 99
Number of participants with dose limiting toxicities (DLT) (Part 1) | Up to Day 57
Number of participants with dose limiting toxicities (DLT) (Part 2) | Up to Day 99

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kankam, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls